CLINICAL TRIAL: NCT04886063
Title: Open-Label Extension of Studies ATH-1017-AD-0201 and ATH-1017-AD-0202 in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Open Label Study of ATH-1017 for Treatment of Mild to Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: ATH-1017-AD-0203 was terminated after the Ph2/3 parent trial (LIFT-AD; NCT04488419) did not meet its primary endpoint, the GST score.
Sponsor: Athira Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATH-1017-AD-0203
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's; Dementia; ATH-1017; Open Label
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Open label extension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Daily subcutaneous (SC) injection of ATH-1017 - 40mg Dosage
  Interventions: Drug: ATH-1017

INTERVENTIONS:
Drug: ATH-1017 — Daily subcutaneous (SC) injection of ATH-1017 in a pre-filled syringe

SUMMARY:
The objective of this study is to determine the safety and tolerability of fosgonimeton (ATH-1017) in subjects with mild to moderate Alzheimer's disease who completed the 26-week randomized treatment in Study ATH-1017-AD-0201 or Study ATH-1017-AD-0202.

DETAILED DESCRIPTION:
This is a multicenter, seamless, open-label extension (OLEX) study of ATH-1017 treatment in subjects with a clinical diagnosis of mild to moderate Alzheimer's disease who completed 26 weeks treatment in the randomized, placebo-controlled, double-blind studies, ATH-1017-AD-0201 and ATH-1017-AD-0202. This OLEX study will provide additional, longer-term safety and tolerability information on ATH-1017 administration up to 48 months in subjects with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed the Week 26 visit of either of the two blinded parent studies (ATH-1017-AD-0201 or ATH-1017-AD-0202).
* Reliable and capable support person/caregiver who is willing to accept responsibility for supervising the daily treatment or, if required, administering study drug.
* Subject capable of giving signed informed consent, or by a legally acceptable representative.
* Subjects must be in generally good health.
* Male subjects and their partners must agree to continue to use a double-barrier method of contraception during the study, including the follow-up period, unless the partner is not of childbearing potential.

Exclusion Criteria:

* Subject has experienced a serious adverse event during the parent study, which could present an increased safety risk during the open label extension.
* New diagnosis of severe major depressive disorder even without psychotic features.
* Any subject with formalized delusions or hallucinations.
* Significant suicide risk.
* Newly-diagnosed malignant tumor, except for the following conditions that are stable in the judgement of the investigator:

  * Adequately treated squamous and basal cell carcinoma, or squamous and basal cell carcinoma in situ
  * Prostate carcinoma in situ

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester-AD-CARE Program, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reda SM, Setti SE, Berthiaume AA, Wu W, Taylor RW, Johnston JL, Stein LR, Moebius HJ, Church KJ. Fosgonimeton attenuates amyloid-beta toxicity in preclinical models of Alzheimer's disease. Neurotherapeutics. 2024 Jul;21(4):e00350. doi: 10.1016/j.neurot.2024.e00350. Epub 2024 Apr 9. PMID 38599894

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the United States and Australia.
Pre-assignment Details: This was a multicenter, open label extension (OLEX) study of ATH-1017 treatment in participants with mild to moderate Alzheimer's disease (AD) who completed 26 weeks of treatment in the randomized, placebo-controlled, double-blind studies (ATH-1017-AD-0201; LIFT-AD or ATH-1017-AD-0202; ACT-AD).
Groups:
- ATH-1017 40 Milligrams (mg): Participants administered ATH-1017 40 mg via subcutaneous (SC) injection (1 mL pre-filled syringe) once-daily (QD).
  Participants entering ATH-1017-AD-0203 on protocol versions prior to V4 were initially administered ATH-1017 70 mg via subcutaneous (SC) injection (1 mL pre-filled syringe) once-daily (QD). Data are reported for the overall safety population, including those who were previously treated with ATH-1017 70 mg.
Period: Overall Study
Arm/Group | ATH-1017 40 Milligrams (mg)
Started | 423
Completed | 35
Not Completed | 388
Not completed — Adverse Event | 50
Not completed — Lack of Efficacy | 31
Not completed — Withdrawal by Subject | 45
Not completed — Physician Decision | 3
Not completed — Protocol Violation | 3
Not completed — Site closure | 4
Not completed — Nursing home replacement | 3
Not completed — Lost to Follow-up | 5
Not completed — Early study termination or other undetermined reasons | 224
Not completed — >1 reason | 20

BASELINE CHARACTERISTICS:
Arm/Group | ATH-1017 40 Milligrams (mg)
Number analyzed (Participants) | 423
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218
  Male | 205
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 17
  White | 384
  More than one race | 0
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Description - To determine the safety and tolerability of ATH-1017 in subjects with mild to moderate Alzheimer's disease (AD) who completed the 26-week randomized treatment in Study ATH-1017-AD-0201 or Study ATH-1017-AD-0202
Time Frame: Up to 173 weeks (study termination)
Population: Safety population: all participants who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | ATH-1017 40 Milligrams (mg)
Number analyzed (Participants) | 423
Participants
  At least 1 TEAE | 323
  No TEAEs | 100

ADVERSE EVENTS:
Time Frame: Up to 173 weeks; the protocolled 206-week treatment duration ended early due to study termination.
Arm/Group | ATH-1017 40 Milligrams (mg)
All-Cause Mortality (participants affected / at risk) | 4/423
Serious Adverse Events (participants affected / at risk) | 54/423
Other Adverse Events (participants affected / at risk) | 348/423
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATH-1017 40 Milligrams (mg) (N=423)
Anaemia (Blood and lymphatic system disorders) | 1
Monoclonal B-cell lymphocytosis (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Aortic valve incompetence (Cardiac disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Early onset familial Alzheimer's disease (Congenital, familial and genetic disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Oesophageal food impaction (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
COVID-19 (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Respiratory syncytial virus infection (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 3
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seizure (Nervous system disorders) | 3
Metabolic encephalopathy (Nervous system disorders) | 2
Altered state of consciousness (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dementia Alzheimer's type (Nervous system disorders) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Acute psychosis (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATH-1017 40 Milligrams (mg) (N=423)
Injection site reactions (General disorders) | 213 — (high-level term)
COVID-19 (Infections and infestations) | 44
Upper respiratory tract infection (Infections and infestations) | 19
Urinary tract infection (Infections and infestations) | 28
Fall (Injury, poisoning and procedural complications) | 24
Eosinophilia (Blood and lymphatic system disorders) | 20

LIMITATIONS AND CAVEATS:
The study was terminated early, following the completion of the parent study (ATH-1017-AD-0201; LIFT-AD)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT04886063/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT04886063/SAP_001.pdf